CLINICAL TRIAL: NCT03070600
Title: Delivering PrEP in Pregnancy
Brief Title: PrEP Implementation for Mothers in Antenatal Care
Acronym: PrIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenyatta National Hospital (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor, Global Health, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000438; 1R01AI125498 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: HIV Infections; Pregnancy Related
Keywords: PrEP
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: We will select 20 clinics from Western Kenya. Ten clinics will be randomized to universal PrEP and ten to targeted PrEP (Table 2). To ensure balance between study arms in terms of key site characteristics, sites will be categorized on HIV prevalence and ANC volume, and restricted randomization will be used for site (cluster) allocation to intervention and control arms (68).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Universal PrEP Counselling (Active Comparator): All enrolled women receiving antenatal care at facilities assigned to Universal PrEP arm will receive standardized HIV risk counseling and then self-select whether they want to use PrEP.
  Interventions: Other: Universal PrEP Counseling
- Targeted PrEP Clinics (Experimental): All enrolled women receiving antenatal care at facilities assigned to the Targeted PrEP arm will be assessed for HIV-risk prior to receiving targeted PrEP counseling.
  Interventions: Other: Targeted PrEP Counseling

INTERVENTIONS:
Other: Universal PrEP Counseling — Counseling at universal sites, will use a standardized counseling script to state that PrEP is available for women at risk for HIV, explain that HIV prevalence in the region is high, and will note that women with HIV positive partners or who don't know their partner's status may be at risk. Counseling will specify that women may have their own reasons to feel at risk or to want PrEP. Following standardized counseling, women will select PrEP at the same visit or will be allowed to deliberate on the decision and come back at the next visit with a decision. Women will be informed that it is advisable to use PrEP if they know their partner is HIV positive or if they do not know their partner's status and will be encouraged to bring untested partners to clinic if status is unknown.
  Arms: Universal PrEP Counselling
Other: Targeted PrEP Counseling — Following enrollment, the targeted PrEP clinics will provide two inter-related innovations over two ANC visits. In the targeted PrEP clinics, any of the following three criteria can trigger enhanced PrEP counseling. A participant that meets any one of these criteria will receive PrEP counseling during the study visit where the criteria is met:
  1. Risk Score >6 (Risk score includes male partner status known/unknown, syphilis infection, and lifetime number of male partners) or any National AIDS and STI Control Programme (NASCOP) risk factors
  2. participant declines partner self-tests regardless of partner HIV status, and/or
  3. their partner declines self-testing or tests positive.
  Arms: Targeted PrEP Clinics

SUMMARY:
In a region with 15-20% HIV prevalence, an estimated 20% of HIV-uninfected women could have HIV exposures in pregnancy. In a theoretical scenario of perfect PrEP coverage, all women at risk receive PrEP while no women not at HIV risk receive PrEP (Figure 4). With mandatory PrEP given to all women (similar to the approaches used for malaria prophylaxis), all women at risk would be covered but many women not at risk receive unnecessary PrEP. Our premise is that a targeted PrEP model may be closer to perfect coverage than a universal offer/self-select model. Implementing targeted PrEP through strategies that include facilitation of partner testing with self-tests could add HIV prevention benefit by increasing partner HIV diagnosis and treatment similar to the initiation of PrEP among pregnant women. By implementing these strategies and measuring uptake, use, and HIV incidence, we can inform the best health systems model for PrEP delivery in pregnancy.

DETAILED DESCRIPTION:
Women living in regions with high HIV prevalence are at high risk of HIV acquisition in pregnancy and postpartum because they infrequently use condoms, do not know their partner's HIV status, and have biologic changes or changes in their partner's sexual partnerships that increase susceptibility. Oral pre-exposure antiretroviral prophylaxis (PrEP) may be an attractive strategy for HIV prevention in pregnancy/postpartum; however, it is important to ensure PrEP reaches women who are at risk for acquiring HIV during pregnancy while avoiding unnecessary PrEP use during pregnancy. Clinicians and women are using PrEP in pregnancy; in qualitative studies, women, health workers and policy-makers support use of PrEP in pregnancy but advocate for models of PrEP delivery that ensure women at risk receive PrEP while minimizing unnecessary PrEP use in women not at risk. Targeting PrEP to women at greatest risk of HIV may maximize benefits, minimize potential risks, and optimize cost-effectiveness. This cluster-randomized clinical trial (RCT) in 20 Maternal Child Health (MCH) clinics in western Kenya (10 clinics per arm, up to 250 women per clinic, up to 5000 women overall), will compare 2 models of PrEP delivery in pregnancy. Clinics will offer universal availability of PrEP (and women self-select whether to use) or targeted offer of PrEP (i.e., offer to women identified as high risk through a standardized risk assessment and partner self-testing, and then women identified as high-risk select whether to use). Leveraging the pre-existing MCH clinic visit schedule will enable programmatically relevant assessment of PrEP uptake, use, and HIV incidence. The outcome of the study will be a model of PrEP delivery in pregnancy that optimizes effectiveness, safety, and cost-effectiveness. Our team has expertise in maternal-child HIV (John-Stewart, Kinuthia), PrEP clinical trials and implementation science (Baeten, Richardson), partner self-testing (Thirumurthy), economics and qualitative research (Barnabas, O'Malley).

AIM 1a. In a cluster-RCT, compare universal PrEP (offer to all; women self-select PrEP) to targeted PrEP (limit the offer to women identified as high risk through a standardized risk assessment and partner self-testing) for outcomes reflecting the balance of PrEP effectiveness and avoiding unnecessary PrEP exposure to women at low or no risk of HIV: HIV incidence at 9 months postpartum among all women (including those who did and did not receive PrEP) and proportion of women exposed to PrEP.

AIM 1b. To compare trial arms for proportion of women 'appropriately' on PrEP (risk factors), PrEP adherence (drug levels) and duration, partners with known HIV status, partners on ART; infant outcomes (growth, birth outcomes, HIV status).

AIM 2. To estimate the incremental cost-effectiveness of targeted PrEP compared to universal PrEP for women during pregnancy and postpartum, per HIV infection and disability-adjusted life-year (DALY) averted.

AIM 3. To qualitatively assess barriers and facilitators to uptake, adherence, acceptability, and feasibility in universal and targeted PrEP models at the organizational, provider, and individual woman level.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for enrollment will include age ≥15 years
* Pregnant at any gestational age
* Tuberculosis negative
* Plans to reside in area for at least one year postpartum
* Plans to receive postnatal and infant care at the study facility
* Not currently enrolled in any other studies.

Exclusion Criteria:

* HIV+ at time of enrollment

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All participants must be pregnant at time of enrollment.
Enrollment: 4447 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace John-Stewart, MD, PhD, Principal Investigator — University of Washington; Jared Baeten, MD, PhD, Principal Investigator — University of Washington; John Kinuthia, MBChB, MMed, Study Director — Kenyatta National Hospital
Locations (20):
- Kenya (20):
  - Ambira Hospital, Ambira
  - Bondo Subcounty Hospital, Bondo
  - Homabay Teaching and Referral Hospital, Homa Bay
  - Kandiege Subcounty Hospital, Kandege
  - Kendu Bay Subcounty Hospital, Kendu Bay
  - Madiany Subcounty Hospital, Madiany
  - Malanga Subcounty Hospital, Malanga
  - Marindi Subcounty Hospital, Marinde
  - Mbita Subcounty Hospital, Mbita
  - Ndhiwa Subcounty Hospital, Ndhiwa
  - Ober Subcounty Hospital, Ober
  - Ongielo Subcounty Hospital, Ongielo
  - Rachuonyo South Subcounty Hospital, Rachuonyo South
  - Rangwe Subcounty Hospital, Rangwe
  - Rwambwa Subcounty Hospital, Rwambwa
  - Siaya Teaching and Referral Hospital, Siaya
  - Suba Subcounty Hospital, Suba
  - Usigu Subcounty Hospital, Usigu
  - Uyawi Subcounty Hospital, Uyawi
  - Yala Subcounty Hospital, Yala

REFERENCES:
- [Background] Dettinger JC, Kinuthia J, Pintye J, Mwongeli N, Gomez L, Richardson BA, Barnabas R, Wagner AD, O'Malley G, Baeten JM, John-Stewart G. PrEP Implementation for Mothers in Antenatal Care (PrIMA): study protocol of a cluster randomised trial. BMJ Open. 2019 Mar 7;9(3):e025122. doi: 10.1136/bmjopen-2018-025122. PMID 30850409
- [Background] Wagner AD, Kinuthia J, Dettinger J, Mwongeli N, Gomez L, Watoyi S, Drake AL, Abuna F, Pintye J, Ochieng B, Odinga D, John-Stewart G, Baeten JM. Challenges of Discrepant HIV Tests in Pregnant Women in the PrEP era-to Treat or Not to Treat? J Infect Dis. 2021 Feb 3;223(2):234-237. doi: 10.1093/infdis/jiaa343. PMID 32561928
- [Background] Pintye J, Davey DLJ, Wagner AD, John-Stewart G, Baggaley R, Bekker LG, Celum C, Chi BH, Coates TJ, Groves AK, Haberer JE, Heffron R, Kinuthia J, Matthews LT, McIntyre JA, Moodley D, Mofenson LM, Mugo N, Mujugira A, Myer L, Shoptaw S, Stranix-Chibanda L, Baeten JM; PrEP in Pregnancy Working Group. Defining gaps in pre-exposure prophylaxis delivery for pregnant and post-partum women in high-burden settings using an implementation science framework. Lancet HIV. 2020 Aug;7(8):e582-e592. doi: 10.1016/S2352-3018(20)30102-8. PMID 32763221
- [Background] Joseph Davey DL, Pintye J, Baeten JM, Aldrovandi G, Baggaley R, Bekker LG, Celum C, Chi BH, Coates TJ, Haberer JE, Heffron R, Kinuthia J, Matthews LT, McIntyre J, Moodley D, Mofenson LM, Mugo N, Myer L, Mujugira A, Shoptaw S, Stranix-Chibanda L, John-Stewart G; PrEP in Pregnancy Working Group. Emerging evidence from a systematic review of safety of pre-exposure prophylaxis for pregnant and postpartum women: where are we now and where are we heading? J Int AIDS Soc. 2020 Jan;23(1):e25426. doi: 10.1002/jia2.25426. PMID 31912985
- [Result] Dettinger JC, Pintye J, Dollah A, Awuor M, Abuna F, Lagat H, Kohler P, John-Stewart G, O'Malley G, Kinuthia J, Beima-Sofie K. Brief Report: "What Is This PrEP?"-Sources and Accuracy of HIV Pre-Exposure Prophylaxis (PrEP) Awareness Among Adolescent Girls and Young Women Attending Family Planning and Maternal Child Health Clinics in Western Kenya. J Acquir Immune Defic Syndr. 2021 Dec 1;88(4):356-360. doi: 10.1097/QAI.0000000000002782. PMID 34379606
- [Result] Nganga N, Dettinger J, Kinuthia J, Baeten J, John-Stewart G, Gomez L, Marwa M, Ochieng B, Pintye J, Mugwanya K, Mugambi M. Prevalence and correlates of pregnancy self-testing among pregnant women attending antenatal care in western Kenya. PLoS One. 2021 Nov 12;16(11):e0258578. doi: 10.1371/journal.pone.0258578. eCollection 2021. PMID 34767573
- [Result] Escudero JN, Dettinger JC, Pintye J, Kinuthia J, Lagat H, Abuna F, Kohler P, Baeten JM, O'Malley G, John-Stewart GC, Beima-Sofie KM. Community Perceptions About Use of Pre-exposure Prophylaxis Among Adolescent Girls and Young Women in Kenya. J Assoc Nurses AIDS Care. 2020 Nov-Dec;31(6):669-677. doi: 10.1097/JNC.0000000000000191. PMID 32675642
- [Result] Pintye J, O'Malley G, Kinuthia J, Abuna F, Escudero JN, Mugambi M, Awuor M, Dollah A, Dettinger JC, Kohler P, John-Stewart G, Beima-Sofie K. Influences on Early Discontinuation and Persistence of Daily Oral PrEP Use Among Kenyan Adolescent Girls and Young Women: A Qualitative Evaluation From a PrEP Implementation Program. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):e83-e89. doi: 10.1097/QAI.0000000000002587. PMID 33273211
- [Result] Rogers Z, Pintye J, Kinuthia J, O'Malley G, Abuna F, Escudero J, Mugambi M, Awuor M, Dollah A, Dettinger JC, Kohler P, John-Stewart G, Beima-Sofie K. Key influences on the decision to initiate PrEP among adolescent girls and young women within routine maternal child health and family planning clinics in Western Kenya. AIDS Care. 2022 Mar;34(3):363-370. doi: 10.1080/09540121.2021.1981217. Epub 2021 Sep 20. PMID 34543077
- [Derived] Gomez L, Kinuthia J, Abuna F, Baeten JM, Dettinger J, Larsen A, Marwa M, Ngumbau N, Odhiambo B, Omondi P, Stern J, Richardson BA, Watoyi S, John-Stewart G, Pintye J; PrEP Implementation for Mothers in Antenatal Care (PrIMA) Study Team. Prenatal exposure to HIV pre-exposure prophylaxis and birth, growth, and social-emotional developmental outcomes throughout early childhood in Kenya: a prospective cohort study. Lancet Glob Health. 2025 Mar;13(3):e467-e478. doi: 10.1016/S2214-109X(24)00471-6. PMID 40021305
- [Derived] Marwa MM, Larsen A, Abuna F, Dettinger J, Odhiambo B, Watoyi S, Omondi P, Ngumbau N, Gomez L, John-Stewart G, Kinuthia J, Pintye J. Brief Report: HIV Risk Perception and Pre-Exposure Prophylaxis Uptake Among Pregnant Women Offered Pre-Exposure Prophylaxis During Antenatal Care in Kenya. J Acquir Immune Defic Syndr. 2025 Jun 1;99(2):116-122. doi: 10.1097/QAI.0000000000003641. PMID 39885623
- [Derived] Ngumbau NM, Neary J, Wagner AD, Abuna F, Ochieng B, Dettinger JC, Gomez L, Marwa MM, Watoyi S, Nzove E, Pintye J, Baeten JM, Kinuthia J, John-Stewart G. Cofactors of Partner HIV Self-testing and Oral PrEP Acceptance Among Pregnant Women at High Risk of HIV in Kenya. J Acquir Immune Defic Syndr. 2024 Mar 1;95(3):238-245. doi: 10.1097/QAI.0000000000003355. PMID 38408215
- [Derived] Pintye J, Kinuthia J, Abuna F, Anderson PL, Dettinger JC, Gomez L, Haberer JE, Marwa MM, Ngumbau N, Omondi P, Odhiambo B, Stern J, Watoyi S, Baeten JM, John-Stewart G; PrEP Implementation for Mothers in Antenatal Care (PrIMA) Study Team. HIV pre-exposure prophylaxis initiation, persistence, and adherence during pregnancy through the postpartum period. AIDS. 2023 Sep 1;37(11):1725-1737. doi: 10.1097/QAD.0000000000003617. Epub 2023 Jun 6. PMID 37289583
- [Derived] Chen S, Pawelec G, Trompet S, Goldeck D, Mortensen LH, Slagboom PE, Christensen K, Gussekloo J, Kearney P, Buckley BM, Ford I, Jukema JW, Westendorp RGJ, Maier AB. Associations of Cytomegalovirus Infection With All-Cause and Cardiovascular Mortality in Multiple Observational Cohort Studies of Older Adults. J Infect Dis. 2021 Feb 3;223(2):238-246. doi: 10.1093/infdis/jiaa480. PMID 32909605

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment ended on July 31, 2019. At that time 4,447 women had enrolled (consented) into the PrIMA study out of an anticipated 4,500.
Groups:
- Targeted PrEP Clinics: All enrolled women receiving antenatal care at facilities assigned to the Targeted PrEP arm will be assessed for HIV-risk prior to receiving targeted PrEP counseling.
  Targeted PrEP Counseling: Following enrollment, the targeted PrEP clinics will provide two inter-related innovations over two ANC visits. In the targeted PrEP clinics, any of the following three criteria can trigger enhanced PrEP counseling. A participant that meets any one of these criteria will receive PrEP counseling during the study visit where the criteria is met:
  1. Risk Score >6 (Risk score includes male partner status known/unknown, syphilis infection, and lifetime number of male partners) or any National AIDS and STI Control Programme (NASCOP) risk factors
  2. participant declines partner self-tests regardless of partner HIV status, and/or
  3. their partner declines self-testing or tests positive.
Period: Overall Study
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Started | 2250 | 2197
Completed | 2156 | 2032
Not Completed | 94 | 165

BASELINE CHARACTERISTICS:
Population: Enrollment for this study ended on July 31, 2019. At the time that enrollment ended, 4,447 participants had enrolled (consented) into the study out of an anticipated 4,500.
Groups:
- Total: Total of all reporting groups
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics | Total
Number analyzed (Participants) | 2250 | 2197 | 4447
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23.9 [20.7 to 28.2] | 24.1 [21.0 to 28.5] | 24.0 [20.9 to 28.3]
Age, Customized [Count of Participants; unit: Participants]
  <25 years of age | 1307 | 1238 | 2545
  25-35 | 830 | 850 | 1680
  35+ | 112 | 108 | 220
  Age missing | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2250 | 2197 | 4447
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2250 | 2197 | 4447
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 2250 | 2197 | 4447

OUTCOME MEASURES:

1. Primary Outcome: Maternal HIV Incidence
Description: Maternal HIV Incidence
Time Frame: 6 weeks, 6 months, 9 months postpartum
Measure: Number (95% Confidence Interval); unit: incidence/100 Person years
Units Other Than Participants: Person-Time (years)
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 2250 | 2197
Number analyzed (Person-Time (years)) | 2372 | 2266
incidence/100 Person years | 0.38 [0.20 to 0.73] | 0.31 [0.15 to 0.65]

2. Primary Outcome: Appropriate PrEP Decision
Description: Scored 1 for high risk women using PrEP and low risk women not using PrEP; 0 for high risk women NOT on PrEP and low risk women using PrEP
Time Frame: Enrollment to 9 months postpartum, the median gestational age at enrollment was 24 weeks (IQR: 20, 30).
Measure: Count of Participants; unit: Participants
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 2250 | 2197
Participants | 1535 | 1299

3. Secondary Outcome: PrEP Adherence
Description: Sequential dried blood spots, PrEP adherence by DBS dichotomous by pregnancy or postpartum thresholds equivalent to ~7 doses per week (≥650 fmol/punch during pregnancy or ≥950 fmol/punch postpartum) based on the thresholds established by the 2009 IMPAACT directly observed PrEP PK study.
Time Frame: Enrollment to 9 months postpartum
Population: Of the 186 participants sampled for this analyses, 427 DBS samples were analyzed (232 universal arm, 195 targeted arm).
Measure: Number; unit: Samples w/ adherence at ~7dose/week
Units Other Than Participants: DBS Samples
Groups:
- Universal Arm- DBS Samples Selected: Participants in the universal arm who initiated PrEP at any time during the study, with DBS randomly selected for analysis.
- Targeted Arm- DBS Samples Selected: Participants in the targeted arm who initiated PrEP at any time during the study, with DBS randomly selected for analysis.
Arm/Group | Universal Arm- DBS Samples Selected | Targeted Arm- DBS Samples Selected
Number analyzed (Participants) | 100 | 86
Number analyzed (DBS Samples) | 232 | 195
Samples w/ adherence at ~7dose/week | 7 | 9

4. Secondary Outcome: PrEP Duration
Description: Number of months on PrEP
Time Frame: Enrollment to 9 months postpartum, the median gestational age at enrollment was 24 weeks (IQR: 20, 30).
Population: This analysis is restricted to participants who initiated PrEP during the study period.
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Universal Arm- PrEP Initiated: Participants in the Universal Arm that initiated PrEP at any point during the study
- Targeted Arm- PrEP Initiated: Participants in the Targeted Arm that initiated PrEP at any point during the study period
Arm/Group | Universal Arm- PrEP Initiated | Targeted Arm- PrEP Initiated
Number analyzed (Participants) | 397 | 323
months | 8.6 [3.2 to 11.4] | 9.0 [3.8 to 11.9]

5. Secondary Outcome: Partner With Known HIV Status
Description: Participants report of partner's HIV status
Time Frame: At 9 months postpartum
Population: This analysis is restricted to participants who reported having a partner at 9-months postpartum.
Measure: Count of Participants; unit: Participants
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 2155 | 2030
Participants | 1680 | 1648

6. Secondary Outcome: Infant Birthweight
Description: Infant Birthweight
Time Frame: time of delivery
Population: This analysis is restricted to mothers with live born infants with birth weight data available in their clinical records.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 1497 | 1370
kg | 3.5 [3.1 to 3.8] | 3.5 [3.1 to 3.8]

7. Secondary Outcome: Infant Growth
Description: Infant height, weight, and age (Weight-for-Age [WAZ], Height-for-Age [HAZ], Weight-for-Height [WHZ] Z-scores). A Z-score of 0 represents the population mean. Indicators of infant malnutrition are defined as Underweight- WAZ Z-score<-2; Stunting-HAZ Z-Score <-2; Wasting- WHZ Z-Score <-2.
Time Frame: 9 months of age
Population: Length measurements could not be ascertained from all infants
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 1847 | 1659
z-score
  Infant WAZ at 9mo PP | 0.12 [-0.61 to 0.88] | -0.01 [-0.77 to 0.86]
  Infant HAZ at 9mo PP: number analyzed (Participants) | 1777 | 1575
  Infant HAZ at 9mo PP | -0.35 [-1.25 to 0.50] | -0.47 [-1.31 to 0.48]
  Infant WHZ at 9mo PP: number analyzed (Participants) | 1774 | 1586
  Infant WHZ at 9mo PP | 0.42 [-0.48 to 1.37] | 0.29 [-0.59 to 1.26]

8. Secondary Outcome: PrEP Use
Description: PrEP Utilization by participants
Time Frame: Enrollment to 9 months postpartum, the median gestational age at enrollment was 24 weeks (IQR: 20, 30).
Measure: Count of Participants; unit: Participants
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 2250 | 2197
Participants | 397 | 323

9. Secondary Outcome: PrEP Acceptance
Description: PrEP accepted by participants
Time Frame: Enrollment to 9 months postpartum, the median gestational age at enrollment was 24 weeks (IQR: 20, 30).
Measure: Count of Participants; unit: Participants
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 2250 | 2197
Participants | 441 | 387

10. Secondary Outcome: Preterm Birth
Description: Birth <37 weeks gestation
Time Frame: At birth
Population: This analysis is restricted to participants who reported a live birth and had gestational age at birth data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 2205 | 2101
Participants | 506 | 309

11. Other Pre Specified Outcome: PrEP Adherence by Self-report
Description: Any missed doses in the last month reported by participants
Time Frame: Enrollment to 9 months postpartum, the median gestational age at enrollment was 24 weeks (IQR: 20, 30).
Measure: Count of Participants; unit: Participants
Groups:
- Universal Arm- PrEP Initiated; Targeted Arm- PrEP Initiated: This analysis is restricted to participants who initiated PrEP during the study period.
Arm/Group | Universal Arm- PrEP Initiated | Targeted Arm- PrEP Initiated
Number analyzed (Participants) | 390 | 320
Participants | 184 | 120

12. Other Pre Specified Outcome: Partner on ART if HIV Positive
Description: Participant report of partner ART use if partner is HIV positive
Time Frame: Enrollment to 9 months postpartum, the median gestational age at enrollment was 24 weeks (IQR: 20, 30).
Population: This analysis is restricted to participants with a partner known to be living with HIV.
Measure: Count of Participants; unit: Participants
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
Number analyzed (Participants) | 39 | 33
Participants | 37 | 31

ADVERSE EVENTS:
Time Frame: Data on adverse events were monitored and data collected on all adverse events from participants at all study visits or via a phone call to study staff (monthly during antenatal care and 6 weeks, 3 months, 6 months, and 9 months postpartum). The median gestational age at enrollment was 24 weeks (IQR: 20, 30).
Arm/Group | Universal PrEP Counselling | Targeted PrEP Clinics
All-Cause Mortality (participants affected / at risk) | 2/2250 | 2/2197
Serious Adverse Events (participants affected / at risk) | 132/2250 | 118/2197
Other Adverse Events (participants affected / at risk) | 7/2250 | 7/2197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Universal PrEP Counselling (N=2250) | Targeted PrEP Clinics (N=2197)
Infant Death (Pregnancy, puerperium and perinatal conditions) | 51 (51) | 47 (47) — Participant experienced a neonatal or infant death during the study period
Infant Hospitalization (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 3 (3) — Participant experienced an infant hospitalization during the study period
Maternal Hospitalization (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 18 (18) — Participant was hospitalized during the study period
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 8 (8) — Loss of pregnancy before 20 weeks gestational age
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 51 (51) | 41 (41) — Loss of pregnancy after 20 weeks gestational age
Molar Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Universal PrEP Counselling (N=2250) | Targeted PrEP Clinics (N=2197)
Kicked out of home (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)
Experienced violence of abuse (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 4 (4)
Breach of confidentiality (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Suicidal behavior (Psychiatric disorders) | 0 (0) | 1 (1)
Persistent or significant psychosocial distress (Psychiatric disorders) | 3 (3) | 1 (1)
Partner thought participant was HIV positive (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Low HIV incidence limited power of the primary outcome; however, similar HIV incidence in both arms suggest that meaningful differences are unlikely. Changing MoH policies and the COVID-19 pandemic affected study operations. Our observed rates of PrEP adherence and persistence could have been influenced by efforts to optimize study retention, and PrEP adherence relied on self-report, which can overestimate adherence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT03070600/Prot_001.pdf
  • Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03070600/SAP_003.pdf